CLINICAL TRIAL: NCT01290601
Title: A Randomized, Active-control, Double-blind, Double-dummy Study to Evaluate the Efficacy and Safety of Tafenoquine for the Treatment of Plasmodium Vivax in Adults
Brief Title: Study to Evaluate the Efficacy and Safety of Tafenoquine for the Treatment of Plasmodium Vivax in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to meet pre-specified endpoint for the day 28 cure rate
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ study 058; A-12055 (Other: IRB)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Malaria; Plasmodium Vivax
Keywords: malaria; Plasmodium vivax; adults; treatment; tafenoquine
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — tafenoquine; Chloroquine; Primaquine

STUDY DESIGN:
Intervention Model Description: Only if Cohort 1 met specified endpoint criteria would Cohort 2 begin enrollment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Tafenoquine (Experimental): Tafenoquine: 2 capsules (200mg base/capsule for a total of 400mg base) and 4 chloroquine placebo capsules for 2 days, followed by 2 tafenoquine capsules and 2 chloroquine placebo capsules for 1 day, followed by 1 primaquine placebo capsule/day for 14 days.
  Interventions: Drug: Tafenoquine
- Cohort 1-Chloroquine (Active Comparator): Chloroquine (1000 mg chloroquine phosphate) and tafenoquine placebo x 2 day, followed by chloroquine (500 mg chloroquine phosphate) and tafenoquine placebo x 1day, followed by primaquine, 15 mg/day for 14 days.
  Interventions: Drug: Chloroquine + Primaquine
- Cohort 2 Tafenoquine (Experimental): Tafenoquine (600 mg base) and chloroquine placebo x 1d, chloroquine placebo x 2 days, followed by primaquine placebo for 14 days.
  Interventions: Drug: tafenoquine
- Cohort 2 Chloroquine (Active Comparator): Chloroquine (1000 mg chloroquine phosphate) and tafenoquine placebo x 1 day, followed by chloroquine (1000 mg chloroquine phosphate) x 1 day, followed by chloroquine (500 mg chloroquine phosphate) x 1day, followed by primaquine, 15 mg/day for 14 days.
  Interventions: Drug: Chloroquine + Primaquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine: 2 capsules (200mg base/capsule for a total of 400mg base) and 4 chloroquine placebo capsules for 2 days, followed by 2 tafenoquine capsules and 2 chloroquine placebo capsules for 1 day, followed by 1 primaquine placebo capsule/day for 14 days.
  Arms: Cohort 1 Tafenoquine
Drug: Chloroquine + Primaquine — Chloroquine (1000 mg chloroquine phosphate) and tafenoquine placebo x 2 day, followed by chloroquine (500 mg chloroquine phosphate) and tafenoquine placebo x 1day, followed by primaquine, 15 mg/day for 14 days.
  Arms: Cohort 1-Chloroquine
Drug: tafenoquine — Tafenoquine (600 mg base) and chloroquine placebo x 1d, chloroquine placebo x 2 days, followed by primaquine placebo for 14 days.
  Arms: Cohort 2 Tafenoquine
Drug: Chloroquine + Primaquine — Chloroquine (1000 mg chloroquine phosphate) and tafenoquine placebo x 1 day, followed by chloroquine (1000 mg chloroquine phosphate) x 1 day, followed by chloroquine (500 mg chloroquine phosphate) x 1day, followed by primaquine, 15 mg/day for 14 days.
  Arms: Cohort 2 Chloroquine

SUMMARY:
This Phase II study is designed to determine whether a single 600 mg dose or 400mg/day for 3 days of tafenoquine is efficacious, and well tolerated for clearing P. vivax malaria infection (blood schizontocidal and gametocytocidal activity) and preventing P. vivax relapse (hypnozoite eradication). It will also further establish the safety and tolerability of these doses of tafenoquine.

DETAILED DESCRIPTION:
This was a randomized, active-control, double-blind, double-dummy study to be conducted in 2 sequential cohorts. Cohort 1 was randomized 2:1 to receive tafenoquine, 400mg/day for 3 days, or the standard blood schizontocidal dosing regimen of chloroquine (1000mg for 2 days followed by 500mg for 1 day) followed by a standard hypnozoite eradication dosing regimen for primaquine (15mg base per day for 14 days). Cohort 2 was to be randomized 2:1 to receive a single 600mg dose of tafenoquine or the standard blood schizontocidal dosing regimen of chloroquine (1000mg for 2 days followed by 500mg for 1 day) followed by a standard hypnozoite eradication dosing regimen for primaquine (15mg base per day for 14 days).

A planned interim analysis was performed after all subjects in Cohort 1 had completed the day 28 assessment and an Independent Data Monitoring Committee (IDMC) convened to evaluate the efficacy and safety of the tafenoquine dosing regimen (400mg once per day for 3 days) used in Cohort 1. Only if the results from Cohort 1 met pre-defined efficacy and safety criteria was enrollment to begin for Cohort 2. The efficacy criterion for achieving the primary endpoint was that the lower limit of the one-sided 95% confidence interval was no less than 85%, and for safety that a review of trends in all AEs, tolerability, medical observations, methemoglobin and other lab data for all subjects indicated the dose was well tolerated.

During the IDMC review it was determined that Cohort 1 failed to meet the pre-specified endpoint for the day 28 cure rate and therefore Cohort 2 should not be initiated and follow-up in Cohort 1 should be completed according to protocol. Following last subject last visit for Cohort 1 the study was terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Positive smear for P. vivax.
2. Parasite density > 500 and < 200,000/μl
3. Age: 20-60 years old
4. Willing to sign consent form
5. Willing to be hospitalized for 29 days and remain in a malaria free region for 60 days thereafter for follow-up.
6. A female is eligible to enter and participate in this study if she is of:

a non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is post-menopausal or, b child-bearing potential, has a negative pregnancy (urine or serum) test at screen, and agrees to comply with recognized contraceptive methods during the treatment stage of the study and for a period of 12 weeks after stopping study drug. Recognized contraceptive methods include, abstinence, implants of levonorgestrel, injectable progestogen, or appropriate double barrier methods using licensed contraceptives such as diaphragm and condom (by the partner) or intrauterine device and condom. The use of oral/patch contraceptives during the study is not considered sufficient contraceptive protection.

Exclusion Criteria:

1. Mixed malaria infections by Field's stain.
2. Female subjects who are pregnant, lactating or unwilling/unable to comply with recognized contraceptive methods during the treatment stage of the study and for a period of 12 weeks after stopping study drug.
3. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
4. Demonstrated glucose-6-phosphate dehydrogenase deficiency.
5. Subject has taken other anti-malarials (mefloquine, primaquine, chloroquine) within the past 30 days by history
6. Clinically significant illness (intercurrent illness e.g. pneumonia, pre-existing condition e.g. renal disease, malignancy or conditions that may affect absorption of study medication e.g. severe diarrhea or any signs of malnutrition as defined clinically).
7. Clinically significant abnormal laboratory values as determined by history, physical examination or routine blood chemistries and hematology values (laboratory guideline values for exclusion are hemoglobin <7 gm/dL, platelets < 50,000/μl, White Blood Cell count (WBC) < 2000/μl, serum creatinine >2.0mg/dL, or ALT or AST more than 3 times the upper limit of normal for age.
8. History of allergy to chloroquine, mefloquine, tafenoquine, primaquine or any other 8-aminoquinolines.
9. Subject has taken another investigational drug within 30 days or 5 half lives (whichever is longer), of study start.
10. History of previous eye surgery or have evidence of corneal or retinal abnormalities identified in baseline ophthalmological examination.
11. Subjects taking concomitant medications likely to affect renal or ophthalmic function or that are known to be metabolized primarily by the cytochrome P450 isoforms 3A4/5 and 2C9 and whose therapeutic effect occurs within a narrow plasma concentration range (e.g. warfarin, ketoconazole).
12. Subjects whom, after examination by the study ophthalmologist, are judged to be at risk for acute angle closure glaucoma.
13. Females who are pre-menarchal.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-09-15; Primary Completion 2005-01-10 (Actual); Study Completion 2005-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sornchai Looaree Suwan, MD, Principal Investigator — Mahidol University
Locations (1):
- Bangkok Hospital for Tropical Diseases/Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warrasak S, Euswas A, Fukuda MM, Ittiverakul M, Miller RS, Krudsood S, Ohrt C. Comparative ophthalmic assessment of patients receiving tafenoquine or chloroquine/primaquine in a randomized clinical trial for Plasmodium vivax malaria radical cure. Int Ophthalmol. 2019 Aug;39(8):1767-1782. doi: 10.1007/s10792-018-1003-2. Epub 2018 Sep 29. PMID 30269312
- [Derived] Fukuda MM, Krudsood S, Mohamed K, Green JA, Warrasak S, Noedl H, Euswas A, Ittiverakul M, Buathong N, Sriwichai S, Miller RS, Ohrt C. A randomized, double-blind, active-control trial to evaluate the efficacy and safety of a three day course of tafenoquine monotherapy for the treatment of Plasmodium vivax malaria. PLoS One. 2017 Nov 9;12(11):e0187376. doi: 10.1371/journal.pone.0187376. eCollection 2017. PMID 29121061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 subjects were randomized and hospitalized at the Bangkok Hospital for Tropical Diseases for the first 29 days of the study and asked to remain in a malaria non-endemic area until 90 days after study start. Subs had f/u's at D60 and D90, and were contacted at D120 for follow-up blood smear. Subjects remained in the study for 121 days.
Pre-assignment Details: During the IDMC review it was determined that Cohort 1 failed to meet the pre-specified endpoint for the day 28 cure rate and therefore Cohort 2 should not be initiated and follow-up in Cohort 1 should be completed according to protocol. Following last subject last visit for Cohort 1 the study was terminated.
Period: Overall Study
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine | Cohort 2 Tafenoquine | Cohort 2 Chloroquine
Started | 46 | 24 | 0 | 0
Completed | 35 | 19 | 0 | 0
Not Completed | 11 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 7 | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine | Total
Number analyzed (Participants) | 46 | 24 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (6.37) | 29.7 (8.57) | 29.7 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 37 | 20 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Oriental | 46 | 24 | 70
Region of Enrollment [Number; unit: participants]
  Thailand | 46 | 24 | 70

OUTCOME MEASURES:

1. Primary Outcome: Adequate Clinical Response (ACR) of Tafenoquine: 28 Day Cure Rate
Description: A subject will be considered a success (cure) if they have an Adequate Clinical Response (ACR). Tafenoquine was efficacious if the lower bound of the two-sided 90% confidence interval for the day 28 cure rate was not less than 85%
Time Frame: 28 Days
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
Number analyzed (Participants) | 46 | 24
Participants
  Adequate Clinical Response (ACR) | 40 | 22
  Early Treatment Failure | 5 | 0
  Late Treatment Failure | 1 | 2

2. Secondary Outcome: Number of Subjects Without Relapse of P. Vivax
Description: Number of subjects without relapse of P. vivax at 2, 3 and 4 months
  - Blood smears were obtained at Days 28, 60, 90 and 120 to confirm the continued absence of P. vivax parasitemia
Time Frame: Day 28, Months 2, 3 and 4
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
Number analyzed (Participants) | 46 | 24
participants
  Cleared at Day 28 | 40 | 22
  Relapsed by Day 60 | 0 | 0
  Relapsed by Day 90 | 0 | 1
  Relapsed by Day 120 | 0 | 1
  Without Relapse by Day 120 | 35 | 19
  Unevaluable by Day 120 | 5 | 2

3. Secondary Outcome: Safety and Tolerability of Tafenoquine as Defined by Most Common Adverse Events (AEs)
Description: To evaluate the safety and tolerability of the tafenoquine dosing regimens as defined by the most common AE's overall, occurring in >10% of subjects in either treatment group
Time Frame: 90 Days
Measure: Number; unit: AEs
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
Number analyzed (Participants) | 46 | 24
AEs
  Blood methemoglobin present | 46 | 22
  Headache | 14 | 4
  Keratopathy | 14 | 0
  Upper respiratory tract infection | 13 | 5
  Dizziness | 12 | 3
  Retinopathy | 9 | 1
  Eosinophilia | 8 | 7
  Abdominal pain | 6 | 5
  Nausea | 6 | 3
  Thrombocytopenia | 6 | 0
  Eosinophil count increased | 5 | 3
  Pyrexia | 5 | 3

4. Secondary Outcome: Parasite and Gametocyte Clearance Time (PCT and GCT)
Description: Serial blood smears to detect the presence of P. vivax parasites and gametocytes, conducted every 12 hours up to and including day 7, until blood smear became negative were utilized to determine the time to clearance. PCT and GCT were considered cleared if 2 consecutive blood smears were negative.
Time Frame: up to day 7 after baseline smear
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
Number analyzed (Participants) | 46 | 24
Hours
  Parasite Clearance Time | 83.4 (31.85) | 40.0 (15.69)
  Gametocyte Clearance Time | 48.3 (33.27) | 22.7 (16.44)

5. Other Pre Specified Outcome: Fever Clearance Time (FCT)
Description: Measure of body temperature every 12 hours through day 7 was used to determine the time (to nearest 12 hours) from initiation of treatment until subjects temperature decreased to 37.2C and remained at or below that level for a minimum of 24 hours.
Time Frame: through day 7
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
Number analyzed (Participants) | 46 | 24
Hours | 41.5 (30.61) | 24.7 (17.69)

ADVERSE EVENTS:
Time Frame: 0 - 90 days
Description: This study was terminated following completion of Cohort 1, and no subjects were enrolled into Cohort 2. Safety results are therefore presented for Cohort 1 only.
Arm/Group | Cohort 1 Tafenoquine | Cohort 1-Chloroquine
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/24
Serious Adverse Events (participants affected / at risk) | 5/46 | 0/24
Other Adverse Events (participants affected / at risk) | 46/46 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Tafenoquine (N=46) | Cohort 1-Chloroquine (N=24)
Acquired methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood methaemoglobin present (Investigations) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Tafenoquine (N=46) | Cohort 1-Chloroquine (N=24)
Eosinophilia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acquired methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Keratopathy (Eye disorders) | 14 (14) | 0 (0)
Retinopathy (Eye disorders) | 9 (9) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aphthous atomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulcerations (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericoronitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Asthenia (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Inflammation localised (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 5 (5)
Infection subcutaneous abscess (Infections and infestations) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Parasitic infection intestinal (Infections and infestations) | 0 (0) | 2 (2)
Plasmodium falciparum infection (Infections and infestations) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 1 (1) | 0 (0)
Nematodiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood methaemoglobin present (Investigations) | 22 (22) | 0 (0)
Eosinophil count increased (Investigations) | 5 (5) | 3 (3)
Hepatic enzyme abnormal (Investigations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Band neutrophil count increased (Investigations) | 1 (1) | 1 (1)
Blast cell count increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (14) | 4 (4)
Dizziness (Nervous system disorders) | 12 (12) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
IDMC determined that Cohort 1 failed to meet specified endpoint for d28 cure rate; Cohort 2 wasn't initiated and follow-up in Cohort 1 should be completed according to protocol. Following last subjects last visit for Cohort 1 study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No